CLINICAL TRIAL: NCT04305938
Title: A Human Clinical Study to Collect Calibration and Performance Data for the RBA-1 and KBS-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kaligia Biosciences, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: KBS004
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Calibration and Validation of Analyte Testing System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Minimally invasive and non-invasive blood analyte measurement — Rapid point-of-care minimally invasive blood analyzer consisting of a spectrometer and a computer loaded with Kaligia software that controls the data acquisition and signal processing to interpret blood analyte measurement.

SUMMARY:
The purpose of the Kaligia Biosciences KBS Systems 1.0(b) analyte monitoring device is to measure the blood analyte levels in patients. The KBS Systems 1.0(b) device avoids the common practice of accessing the vein to draw blood for conventional laboratory analysis. Instead, the KBS Systems 1.0(b) device uses Raman Spectroscopy to acheive the measurement of various blood analytes through the use of only approximately 40µl of blood. Such a small volume of blood can be sampled via a finger prick procedure rather than needing a larger volume of blood sampled via a venipuncture. The spectra contain information of all the molecules present in the blood (RBCs, hemoglobin, glucose, sodium, potassium, etc.). From these spectra, the system is able to analyze the blood and provide results in a matter of minutes, rather than hours or even, in some cases, days.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 yrs of age.
* Willingness and ability to provide informed consent
* Hospital patients with a physician-prescribed laboratory blood test

Exclusion Criteria:

1. People with clotting factor disorders and/or currently taking anticoagulation medication.
2. Has any other medical condition that, in the opinion of the Investigator, would interfere with the person's participation in this study (i.e. double arm amputee).
3. Any skin abnormalities or tattoos located on the palm(s) of the hand(s). The left palm is preferred for this study; however, the right palm can be used if the left palm is excluded.
4. Parkinson's disease, dyskinesia, tremors, or similar that may make it challenging for said person to hold their hand on the device in a still and stable manner.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The research subjects subjected to the test articles used in this study will be hospital patients with doctor-prescribed blood tests as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Analyte validation | 6 months
  CLIA laboratory analyte values will be compared to device analyte readings and inform machine learning of device software learning to achieve device calibration and validation of readings.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided